CLINICAL TRIAL: NCT07052032
Title: A Phase 1b, Open-Label, Multicenter Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, Immunogenicity, and Preliminary Clinical Activity of CND261 in Patients With Seropositive Rheumatoid Arthritis
Brief Title: An Open-label Study of CND261 in Seropositive Rheumatoid Arthritis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Candid Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CND261-101
Record Dates: First submitted 2025-06-18; First posted 2025-07-04 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CND261 (Experimental)
  Interventions: Biological: CND261

INTERVENTIONS:
Biological: CND261 — CND261 will be dosed according to the assigned cohort

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of CND261 in patients with seropositive rheumatoid arthritis.

DETAILED DESCRIPTION:
This is a Phase 1b, open-label, multicenter study evaluating the safety, tolerability, pharmacokinetics, pharmacodynamics, immunogenicity, and preliminary clinical activity of CND261 in patients with seropositive rheumatoid arthritis. The study consists of 2 parts: a dose-escalation part and an open-label expansion. Patients will be followed until Week 52.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 75 years old
2. Diagnosis of adult-onset RA
3. Class I-III RA
4. Moderately to severely active RA
5. Inadequate treatment response as defined in the protocol
6. Stable use of any concomitant therapies

Exclusion Criteria:

1. Inadequate clinical laboratory parameters at Screening
2. Active infection
3. Receipt of or inability to discontinue any excluded therapies
4. Receipt of live vaccine within 4 weeks
5. Presence of any concomitant autoimmune disease
6. Active or known history of catastrophic anti-phospholipid syndrome
7. APS or thrombotic event not adequately controlled by anticoagulation therapy
8. History of progressive multifocal leukoencephalopathy
9. Central nervous system disease
10. Presence of 1 or more significant concurrent medical conditions
11. Have a diagnosis or history of malignant disease within 5 years
12. Serious mental illness, alcohol or drug abuse, dementia, or any other condition that would impair ability to receive planned treatment or to understand informed consent
13. History of or planned organ transplant and/or autologous or allogeneic hematopoietic stem cell transplantation
14. Major surgery requiring use of general anesthesia within 12 weeks or planned or expected major surgery during the study
15. Women who are pregnant or breastfeeding
16. Patients who do not agree to the use of highly effective contraception as defined by the protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events through end of study | Baseline to Month 12
Changes from baseline in vital signs through end of study | Baseline to Month 12
Changes from baseline in ECG parameters through end of study: PR interval | Baseline to Month 12
Changes from baseline in ECG parameters through end of study: QRS interval | Baseline to Month 12
Changes from baseline in ECG parameters through end of study: QTcF interval | Baseline to Month 12
Changes from baseline in safety laboratory assessments through end of study | Baseline to Month 12

SECONDARY OUTCOMES:
Pharmacokinetic (PK) concentration-time profiles for CND261 | Baseline to Month 12
PK parameters for CND261: maximum concentration | Baseline to Month 12
PK parameters for CND261: time of maximum concentration | Baseline to Month 12
PK parameters for CND261: area under the concentration-time curve | Baseline to Month 12
PK parameters for CND261: clearance | Baseline to Month 12
PK parameters for CND261: volume of distribution | Baseline to Month 12
PK parameters for CND261: half-life | Baseline to Month 12

CONTACTS AND LOCATIONS:
Locations (6):
- Candid Clinical Site, Tbilisi, Georgia
- Candid Clinical Site, Chisinau, Moldova
- Candid Clinical Site, Auckland, New Zealand
- Romania (2):
  - Candid Clinical Site, Bucharest
  - Candid Clinical Site, Cluj-Napoca
- Candid Clinical Site, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: No